CLINICAL TRIAL: NCT04644029
Title: A Phase 3, Randomized, Active-Controlled, Double-blind Clinical Study to Evaluate the Efficacy and Safety of Oral Islatravir Once-Monthly as Preexposure Prophylaxis in Cisgender Women at High Risk for HIV-1 Infection
Brief Title: Oral ISL QM as PrEP in Cisgender Women at High Risk for HIV-1 Infection (MK-8591-022)
Acronym: Impower-022
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Voluntarily terminated due to benefit/risk assessment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 8591-022; MK-8591-022 (Other: Merck); 2021-001289-39 (EudraCT Number)
Record Dates: First submitted 2020-11-23; First posted 2020-11-25 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: HIV-I; Human Immunodeficiency Virus Type 1; Prophylaxis
Keywords: Preexposure prophylaxis (PrEP); Prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — islatravir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: In Study Part 1, a double-blinding technique with in-house blinding will be used. ISL and FTC/TDF will be packaged identically relative to their matching placebos so that blind is maintained. The participant, the investigator, and Sponsor personnel or delegate(s) who are involved in the study intervention administration or clinical evaluation of the participants are unaware of the intervention assignments.
  In Study Part 2, sponsor personnel not directly involved with blinded safety monitoring will be unblinded to participants' randomized study intervention in Part 1.
  In Study Part 3, participants, investigators, and all Sponsor personnel will be unblinded to the participants' original randomized study intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ISL QM (Experimental): ISL (islatravir) once monthly AND placebo to FTC/TDF (emtricitabine/tenofovir disoproxil) once daily. Following study-wide cessation of ISL administration, participants had the option to receive open-label FTC/TDF administered once daily.
  Interventions: Drug: Islatravir; Drug: Placebo to FTC/TDF
- FTC/TDF QD (Active Comparator): FTC/TDF (TRUVADA™ or generic product emtricitabine/tenofovir disoproxil) administered once daily. Placebo to ISL (islatravir) administered once monthly. Following study-wide cessation of ISL administration, participants had the option to continue on open-label FTC/TDF. Placebo was no longer administered once open label treatment began.
  Interventions: Drug: FTC/TDF; Drug: Placebo to ISL

INTERVENTIONS:
Drug: Islatravir — Oral 60 mg tablet administered once monthly during Part 1.
  Other Names: MK-8591
  Arms: ISL QM
Drug: Placebo to FTC/TDF — 0 mg tablet administered once daily during Part 1.
  Arms: ISL QM
Drug: FTC/TDF — Each tablet contains 200 mg emtricitabine and 245 mg of tenofovir disoproxil (equivalent to 300 mg tenofovir disoproxil fumarate or 201.22 mg tenofovir disproxil phosphate), administered orally once daily in Parts 1, 2, and 3.
  Other Names: TRUVADA™; Emtricitabine/Tenofovir disoproxil; Emtricitabine/Tenofovir disoproxil fumarate
  Arms: FTC/TDF QD
Drug: Placebo to ISL — 0 mg tablet administered orally once monthly in Part 1.
  Arms: FTC/TDF QD

SUMMARY:
This study will evaluate whether oral islatravir (ISL) is effective in preventing Human Immunodeficiency Virus Type 1 (HIV-1) infection in women at high-risk for HIV-1 infection. The study will compare oral ISL taken once a month with standard-of-care medication for prevention of HIV-1 infection, emtricitabine/tenofovir disoproxil (FTC/TDF), taken once per day. The primary hypothesis is that oral ISL is more effective than FTC/TDF at reducing the incidence rate per year of confirmed HIV-1 infections.

DETAILED DESCRIPTION:
Based on laboratory findings of decreased lymphocyte and CD4+ T-cell counts across the islatravir program, dosing of blinded study intervention was halted on 13-Dec-2021 and screening and randomization of new participants was ended. Blinded assessments conducted prior to this date are designated as Study Part 1. During Study Part 2, participants from Part 1 have the option to receive daily open-label FTC/TDF while continuing in the study for safety monitoring. Study Part 3 was added to unblind each participant's Part 1 study intervention assignment, continue participants on FTC/TDF, and monitor safety.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-uninfected based on negative HIV-1/HIV-2 test results before randomization.
* Sexually active (vaginal and/or anal sex) with a male sexual partner in the 30 days prior to screening.
* High risk for HIV-1 infection.
* Not pregnant or breastfeeding, and one of the following conditions applies: Not a woman of childbearing potential (WOCBP) or is a WOCBP and is using an acceptable contraceptive method during the intervention period and for at least 42 days after the last dose.
* A WOCBP must have a negative pregnancy test within 24 hours prior to the first dose of study intervention.

Exclusion Criteria:

* Hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator.
* Findings of chronic hepatitis B virus (HBV) infection or past HBV.
* Current or chronic history of liver disease.
* History of malignancy within 5 years of screening except for adequately-treated basal cell or squamous cell skin cancer, or in situ cervical cancer.
* Past or current use of cabotegravir, lenacapavir, or any other long-acting HIV prevention product.
* Currently participating in or has participated in an interventional clinical study with an investigational compound or device, within 30 days prior to Day 1.
* Expecting to conceive or donate eggs at any time during the study.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Assigned female sex at birth and is cisgender
Enrollment: 730 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (24):
- United States (13):
  - University of Alabama at Birmingham-UAB Sexual Health Research Clinic (SHRC) ( Site 0064), Birmingham, Alabama
  - MedStar Health Research Institute (MedStar Physician Based R-MedStar Washington Hospital Center ( Si, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine-Infectious Disease ( Site 0076), Miami, Florida
  - Orlando Immunology Center ( Site 0068), Orlando, Florida
  - Ponce De Leon Center Grady Health ( Site 0066), Atlanta, Georgia
  - The University of Mississippi Medical Center ( Site 0065), Jackson, Mississippi
  - KC CARE Health Center-Clinical Trials ( Site 0059), Kansas City, Missouri
  - Rutgers New Jersey Medical School-Clinical Research Center ( Site 0071), Newark, New Jersey
  - Bronx Prevention Center ICAP ( Site 0062), The Bronx, New York
  - The University of North Carolina at Chapel Hill-Medicine ( Site 0056), Chapel Hill, North Carolina
  - Prisma Health Richland Hospital-Clinical Research Unit ( Site 0069), Columbia, South Carolina
  - Prism Health North Texas, Oak Cliff Health Center ( Site 0070), Dallas, Texas
  - West Virginia University-Department of Medicine ( Site 0061), Morgantown, West Virginia
- South Africa (10):
  - Perinatal HIV Research Unit (PHRU)-HIV Prevention CRS ( Site 0023), Johannesburg, Gauteng
  - Wits Reproductive Health and HIV Institute (WRHI)-Wits RHI Ward 21 Clinical Research site ( Site 002, Johannesburg, Gauteng
  - Helen Joseph Hospital-Clinical HIV Research Unit ( Site 0020), Johannesburg, Gauteng
  - Setshaba Research Centre ( Site 0016), Pretoria, Gauteng
  - SA Medical Research Council - Chatsworth Clinical Research Site ( Site 0030), Chatsworth, KwaZulu-Natal
  - Maternal Adolescent and Child Health Research (MatCH) ( Site 0025), Durban, KwaZulu-Natal
  - Qhakaza Mbokodo Research Clinic ( Site 0017), Ladysmith, KwaZulu-Natal
  - Madibeng Centre for Research ( Site 0019), Brits, North West
  - Aurum Institute Klerksdorp CRS ( Site 0029), Klerksdorp, North West
  - Aurum Institute - Rustenburg ( Site 0022), Rustenburg, North West
- MU-JHU Care Limited-Clinic ( Site 0041), Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26659&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One person mistakenly received study drug without being randomized. They are not included in Participant Flow or Baseline Characteristics because they were not enrolled in the study, but their adverse events are reported in the Adverse Events module because they received study drug.
Groups:
- ISL QM: ISL (islatravir) once monthly AND placebo to FTC/TDF (emtricitabine/tenofovir disoproxil) once daily. Following study-wide cessation of ISL administration, participants had the option to receive open-label FTC/TDF. Placebo was no longer administered once open label treatment began.
Period: Overall Study
Arm/Group | ISL QM | FTC/TDF QD
Started | 364 | 366
Treated Per Protocol Arm Design | 362 | 365
Received Open-Label FTC/TDF | 343 | 345
Completed | 0 | 0
Not Completed | 364 | 366
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 21 | 19
Not completed — Lost to Follow-up | 31 | 34
Not completed — Study Terminated by Sponsor | 308 | 309
Not completed — Randomized in Error | 2 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline characteristics population includes all randomized participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | ISL QM | FTC/TDF QD | Total
Number analyzed (Participants) | 362 | 365 | 727
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.0 (6.1) | 26.1 (6.3) | 26.1 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 362 | 365 | 727
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 24
  Not Hispanic or Latino | 329 | 330 | 659
  Unknown or Not Reported | 22 | 22 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 334 | 338 | 672
  White | 19 | 15 | 34
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate Per Year of Confirmed HIV-1 Infection Among Participants During Blinded Treatment +42 Days Post-Blind
Description: Incidence rate per year of confirmed HIV-1 infections is the number of participants with confirmed HIV-1 infections during the assessment period divided by the number of person-years in the arm. Data are based on participants with confirmed HIV-1 infection. The originally planned primary statistical analysis was removed via amendment when open-label treatment was initiated.
Time Frame: Up to approximately 325 days
Population: The analysis population includes all participants who were randomized and received at least 1 dose of study intervention and did not have confirmed HIV-1 infections prior to or at randomization.
Measure: Number; unit: Percentage of Participants/Person-Year
Arm/Group | ISL QM | FTC/TDF QD
Number analyzed (Participants) | 362 | 363
Percentage of Participants/Person-Year | 0.000 | 0.000

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE) During Blinded Treatment + 42 Days Post-Blind
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced an AE will be reported for each treatment arm.
Time Frame: Up to approximately 325 days
Population: The analysis population includes all participants who were randomized and received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | ISL QM | FTC/TDF QD
Number analyzed (Participants) | 362 | 365
Participants | 198 | 255

3. Primary Outcome: Number of Participants Who Discontinued Blinded Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued blinded study treatment due to an AE will be reported for each treatment arm.
Time Frame: Up to 283 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ISL QM | FTC/TDF QD
Number analyzed (Participants) | 362 | 365
Participants | 2 | 4

4. Secondary Outcome: Incidence Rate Per Year During Blinded Treatment of Confirmed HIV-1 Infection Among ISL-Treated Participants
Description: Incidence rate per year of confirmed HIV-1 infections is the number of participants with confirmed HIV-1 infections during the assessment period divided by the number of person-years in the arm. Data are based on participants with confirmed HIV-1 infection. The originally planned secondary statistical analysis was removed via amendment when open-label treatment was initiated.
Time Frame: Up to approximately 237 days
Population: The analysis population includes all participants who were randomized and received at least 1 dose of ISL and did not have confirmed HIV-1 infections prior to or at randomization.
Measure: Number; unit: Percentage of Participants/Person-Year
Arm/Group | ISL QM
Number analyzed (Participants) | 362
Percentage of Participants/Person-Year | 0.000

ADVERSE EVENTS:
Time Frame: Blinded arms and mistaken treatment arm: Up to approximately 325 days Open-label arms: Up to approximately 639 days (starting 42 days after last blinded treatment; includes the time leading up to first open-label treatment)
Description: Following sponsor decision to stop dosing blinded study treatment, all participants were offered the option to receive open-label FTC/TDF. Open-label treatment arms include all events occurring more than 42 days after a participant's final blinded treatment, even if those events occurred prior to their first open-label treatment.
  AEs are presented for all randomized-and-treated participants. All-Cause Mortality includes all randomized participants starting from the time of randomization.
Groups:
- ISL QM: ISL (islatravir) once monthly AND placebo to FTC/TDF (emtricitabine/tenofovir disoproxil) once daily. Following study-wide cessation of ISL administration, participants had the option to receive open-label FTC/TDF administered once daily. Adverse events during the open-label period are not counted in this arm.
- ISL QM > Open-Label FTC/TDF: This arm represents participants who received open-label FTC/TDF (TRUVADA™ or generic product emtricitabine/tenofovir disoproxil) administered once daily, after previously receiving ISL QM during the blinded portion of the study.
- FTC/TDF QD: FTC/TDF (TRUVADA™ or generic product emtricitabine/tenofovir disoproxil) administered once daily. Placebo to ISL (islatravir) administered once monthly. Following study-wide cessation of ISL administration, participants had the option to continue on open-label FTC/TDF. Placebo was no longer administered once open label treatment began. Adverse events during the open-label period are not counted in this arm.
- FTC/TDF > Open-Label FTC/TDF Second Course: This arm represents participants who received open-label FTC/TDF (TRUVADA™ or generic product emtricitabine/tenofovir disoproxil) administered once daily, after previously receiving FTC/TDF QD during the blinded portion of the study.
- FTC/TDF-Treated Without Randomization: The participant in this arm was mistakenly given daily FTC/TDF plus monthly placebo to ISL without completing enrollment and randomization. Following study unblinding, participant continued to receive open-label daily FTC/TDF. Adverse events were collected for this participant during blinded and open-label treatment due to receiving study drug, but zero participants are reported as affected and zero adverse event instances are reported due to the risk of identification of a person.
Arm/Group | ISL QM | ISL QM > Open-Label FTC/TDF | FTC/TDF QD | FTC/TDF > Open-Label FTC/TDF Second Course | FTC/TDF-Treated Without Randomization
All-Cause Mortality (participants affected / at risk) | 1/364 | 0/343 | 0/366 | 0/345 | 0/1
Serious Adverse Events (participants affected / at risk) | 4/362 | 13/343 | 2/365 | 23/345 | 0/1
Other Adverse Events (participants affected / at risk) | 145/362 | 292/343 | 210/365 | 284/345 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISL QM (N=362) | ISL QM > Open-Label FTC/TDF (N=343) | FTC/TDF QD (N=365) | FTC/TDF > Open-Label FTC/TDF Second Course (N=345) | FTC/TDF-Treated Without Randomization (N=1)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crush injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failed trial of labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Spontaneous rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISL QM (N=362) | ISL QM > Open-Label FTC/TDF (N=343) | FTC/TDF QD (N=365) | FTC/TDF > Open-Label FTC/TDF Second Course (N=345) | FTC/TDF-Treated Without Randomization (N=1)
Diarrhoea (Gastrointestinal disorders) | 19 (19) | 14 (16) | 29 (32) | 21 (23) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (21) | 13 (16) | 41 (43) | 13 (15) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (9) | 15 (17) | 22 (25) | 12 (13) | 0 (0)
Fatigue (General disorders) | 10 (12) | 5 (8) | 19 (19) | 5 (5) | 0 (0)
Influenza like illness (General disorders) | 4 (4) | 45 (65) | 3 (3) | 41 (62) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 28 (30) | 158 (263) | 57 (59) | 143 (255) | 0 (0)
Chlamydial infection (Infections and infestations) | 4 (4) | 58 (78) | 17 (17) | 55 (71) | 0 (0)
Gastroenteritis (Infections and infestations) | 7 (7) | 16 (18) | 6 (6) | 18 (18) | 0 (0)
Trichomoniasis (Infections and infestations) | 2 (2) | 28 (36) | 11 (12) | 24 (28) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 21 (24) | 70 (89) | 12 (13) | 55 (74) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 31 (38) | 5 (5) | 34 (38) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 13 (13) | 114 (163) | 29 (30) | 109 (160) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 17 (22) | 1 (1) | 21 (25) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 19 (20) | 3 (3) | 10 (11) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 21 (28) | 4 (5) | 18 (21) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 4 (4) | 18 (24) | 4 (4) | 14 (18) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 26 (36) | 4 (4) | 20 (32) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 16 (19) | 8 (8) | 25 (28) | 0 (0)
Dizziness (Nervous system disorders) | 17 (17) | 11 (12) | 27 (28) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 43 (50) | 61 (90) | 53 (65) | 56 (83) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 13 (16) | 33 (42) | 11 (15) | 39 (53) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 7 (7) | 30 (36) | 11 (12) | 30 (38) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT04644029/Prot_SAP_001.pdf